CLINICAL TRIAL: NCT01643109
Title: Childhood Hemiplegic CP Integrated Neuroscience Discovery Network (CP-NET) Theme IIIa: Constraint Induced Movement Therapy (CIMT)- Neuroimaging Predictors of Positive Response to Constraint
Brief Title: Constraint Induced Movement Therapy (CIMT)- Neuroimaging Predictors of Positive Response to Constraint
Acronym: OBI_CIMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-294
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Cerebral Palsy; Hemiplegia; Constraint Induced Movement Therapy
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CIMT (Experimental): A standardized CIMT protocol will be administered over a three week period. The first week will consist of wearing a below elbow cast on the non-hemiplegic limb followed by a two week CIMT camp (5 hours per day, 5 days per week) where the child/youth wears a constraint splint on the non-hemiplegic hand. The two week camp will follow a standardized CIMT camp protocol ("Hand2Hand" developed at HBKRH) that includes activities that focus on unilateral hemiplegic hand activity in the first week and increasing incorporation of bilateral hand activities in the second week. The camp protocol for CIMT is based on camp protocols utilized successfully in other paediatric research studies.
  Interventions: Other: Casting & CIMT
- Comparison (No Intervention): Standard therapy.

INTERVENTIONS:
Other: Casting & CIMT — A standardized CIMT protocol will be administered over a three week period. The first week will consist of wearing a below elbow cast on the non-hemiplegic limb followed by a two week CIMT camp (5 hours per day, 5 days per week) where the child/youth wears a constraint splint on the non-hemiplegic hand. The two week camp will follow a standardized CIMT camp protocol ("Hand2Hand" developed at HBKRH) that includes activities that focus on unilateral hemiplegic hand activity in the first week and increasing incorporation of bilateral hand activities in the second week. The camp protocol for CIMT is based on camp protocols utilized successfully in other paediatric research studies.
  Arms: CIMT

SUMMARY:
CIMT has shown great promise in helping children and adults regain lost function in a disabled limb by forcing its use through an intensive motor training program and constraining the unaffected arm with a cast. However, relatively little is known about the underlying mechanisms of CIMT in hemiplegic CP. This project will use an integrated translation model to explore neuroimaging predictors of a positive clinical response to CIMT.

DETAILED DESCRIPTION:
The primary research objective is to evaluate neuroimaging predictors of a positive response to CIMT in children with hemiplegic CP secondary to a middle cerebral artery territory stroke (MCA). A focus on the MCA territory is chosen as (1) it targets children with significant hand impairment who have the potential to benefit from CIMT, (2) is the most common neuropathological subtype, and (3) allows for enhanced homogeneity for the matching of case and comparison groups. The primary research question is: In children aged 7 to 16 years with hemiplegic CP secondary to an MCA stroke, are there neuroimaging predictors of a positive response to CIMT, a positive response being defined by an improvement in the Assisting Hands Assessment (AHA) one month after CIMT?

Neuroimaging predictor variables include laterality index (LI) of the primary M1 and S1 areas on fMRI, IHI evaluated by resting state fMRI, dissociation of the M1 and S1 for the hemiplegic hand measured by fMRI, size and vascular distribution of the MCA lesion with T2 weighted MRI, and white matter tract abnormality with Diffusion Tensor Imaging (DTI). We hypothesize that a negative LI, a non-dissociated M1 and S1, low IHI, small size of infarction, and large size of the contralateral corticospinal tract will predict a positive response to constraint. An evaluation of the neuroimaging predictor variables on the persistence of a positive response to CIMT at 6 months as measured by the AHA will also be explored. A secondary objective will evaluate change in the neuroimaging variables from baseline to one month post CIMT by comparing children in the case group who have received CIMT and a comparison group who are matched on baseline QUEST scores.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hemiplegic CP secondary to an MCA infarct
* Age between 7 and 16 years
* Ability to co-operate, understand, and follow simple instructions for neuro-imaging outcome measurement: The functional MRI protocol will require some cooperation and the child will need to lie still in a confined place for approximately 45-60 min.
* No previous CIMT within 12-months of study entry or Botulinum toxin upper limb injections within 6-months of study entry.

Exclusion Criteria:

* None

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Assisted Hand Assessment | baseline, 1-month after intervention and 6-months
  The primary outcome measure for this study will be the assisted hand assessment (AHA). This test is the gold standard in paediatric constraint research to assess the use of the assisting hand in bilateral activities (hand use) in children with hemiplegic CP with established reliability, validity and responsiveness. Importantly it has undergone the rigour of a Rasch analysis in its development.

CONTACTS AND LOCATIONS:
Overall Officials: Darcy L Fehlings, MD MSc, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (3):
- Canada (3):
  - McMaster Children's Hospital, Hamilton Health Sciences, Hamilton, Ontario
  - Thames Valley Children's Centre, London Health Sciences Centre, London, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario